CLINICAL TRIAL: NCT04097639
Title: An Observational Study Designed to Elucidate the Pathways by Which Low-grade Inflammation Contributes to Anaemia in Rural African Children From 6 Months to 2 Years of Age
Brief Title: Inflammation, Iron Deficiency and Anaemia Study 1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: SCC 1664
Record Dates: First submitted 2019-05-03; First posted 2019-09-20 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Anemia
Keywords: low-grade inflammation; anemia; erythroferrone
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigator have previously shown that hepcidin is up-regulated even by low levels of inflammation and, according to our prior stable isotope studies, is predicted to block iron absorption. In this follow-up observational study, investigator aim to elucidate the potential drivers of this low-grade inflammation and to recalibrate the relationship between hepcidin and iron absorption using a more direct measure of absorption than the stable isotope method which measures the net of absorption and utilization. Investigator will study 120 ostensibly well children (6-24m) living in the rural region of West Kiang.

Investigator will:

1. Use detailed clinical screening for possible origins of the low grade inflammation.
2. Assess iron absorption and its relationship to iron and anaemia status, inflammation, EPO, erythroferrone and hepcidin.

DETAILED DESCRIPTION:
Aim 1:

Hypothesis 1: 'Minor' but persistent infections of the respiratory tract, skin, mouth, and gut cause chronic elevation of hepcidin levels and other markers of infection including CRP.

Research Question 1: What is the relationship between each of the following: CRP, hepcidin, clinical score of skin infections; clinical score of oral health; clinical score of respiratory infections; and systemic markers of gut damage and bacterial translocation (serum EndoCAB and iFABP) and stool markers of inflammation (calprotectin, REG1b and lipocalin2).

Hypothesis 2: Respiratory infections and airway inflammation are the most common cause of low grade inflammation.

Research Question 2: What is the most common source(s) of persistent low-grade inflammation in apparently well children living in rural Gambia.

Aim 2:

Hypothesis: Hepcidin levels above 5.5ng/ml block oral iron absorption.

Research Question: What is the relationship between hepcidin and oral iron absorption in well children living in rural Gambia?

Aim 3:

Hypothesis: Anaemic children with low-grade inflammation have anaemia of inflammation with concomitant iron deficiency that results in inappropriately low levels of EPO production and reticulocytosis for their erythroid mass (Hb levels) levels.

Research Question: Is there decreased EPO synthesis and/or increased EPO resistance in anaemic children with low-grade inflammation living in rural Gambia?

Aim 4:

Hypothesis: First investigator will conduct a hypothesis-free exploratory analysis to assess whether erythroferrone behaves as predicted based upon mouse models (ie up-regulated by stress erythropoiesis and inversely related to hepcidin). Investigator additionally hypothesize that there may be a vicious cycle initiated by inflammation and then perpetuated by the consequent low levels of (iron-restricted) erythropoiesis, leading to low erythroferrone and loss of hepcidin suppression.

Research Question: What is the relationship between erythroferrone, iron status, inflammation, hepcidin, EPO in anaemic and non-anaemic children with and without low-grade inflammation living in rural Gambia? Primary: To examine in detail the pathways by which low-grade inflammation causes iron deficiency anaemia in African children.

Secondary: To assess if anaemia of inflammation and resistance to erythropoietin play a role in causing and perpetuating anaemia in children living in rural Africa.

This is an observational study of 120 children who will be recruited at the routine vaccination clinics or pre-scheduled well-child check-ups at the Keneba clinic. Each child will be seen three times (at 6, 12 and 18 months) and the same protocol will be used at each visit.

Figure 1: Study design At each visit, children will be examined by the Research Clinician or PI using pre-determined validated checklists for possible sources of low-grade inflammation. Each participant will be given a clinical score for skin conditions, oral health, and respiratory infections/airway disease.

After the clinical examination, an oral iron absorption protocol will be initiated:

Step 1: A venous blood sample will be collected and assayed for full blood count (including reticulocyte count) and serum iron markers, hepcidin, erythropoietin (EPO), erythroferrone, IL-6 and EndoCab; Step 2: Children will be given an oral dose of liquid ferrous fumarate at 2mg/kg; Step 3: Between 3-4 hours later a venous blood sample will be drawn for measurement serum iron markers. The change in serum iron levels (measured before and after dosing) will be used as a direct measurement of iron absorption.

ELIGIBILITY:
Inclusion Criteria:

* 1)Male or female children ages 6-8 months at the time of study enrolment.
* 2)Signed or fingerprinted or personally marked written informed consent obtained from their parent/guardian.
* 3)Parent/guardian plans for subject to reside in study site area and are able and willing to adhere to all protocol visits and procedures.

Exclusion Criteria:

* 1) Acute illness
* 2) Fever (for eligibility purpose defined as a body temperature greater than 37.5°C) if appropriate, as per investigator assessment, subject may be re-revaluated for eligibility).
* 3)Vaccination less than 7 days prior to study enrollment.
* 4)Administration of immunosuppressants or other immune-modifying agents within 90 days prior to study IP administration (e.g., systemic corticosteroids at doses equivalent to ≥ 0.5 mg/kg/day of prednisone for more than 14 days; topical steroids including inhaled and intranasal steroids are not exclusionary).
* 5)Administration of systemic antibiotic treatment within 3 days prior to study enrolment.
* 6)Any history of or evidence for chronic clinically significant (as per investigator assessment) disorder or disease (including, but not limited to, immunodeficiency, autoimmunity, malnutrition*, congenital abnormality, bleeding disorder, and pulmonary, cardiovascular, metabolic, neurologic, renal, or hepatic disease).
* 7)Any history of maternal human immunodeficiency virus, chronic hepatitis B or chronic hepatitis C infections.
* 8)Any condition that in the opinion of the investigator might compromise the safety or well-being of the subject or compromise adherence to protocol procedures.
* 9)Participation in another MRC study.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population is young children to who's mothers/guardians the study protocol will be explained orally in the presence of a witness in case they are illiterate or in writing and we will not start any study specific procedure before informed consent is obtained
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Serum hepcidin level | 18 months
  To examine in detail the pathways by which low-grade inflammation causes iron deficiency anaemia in African children
clinical score of site and severity of infection and inflammation | 18 months
  Clinical score of skin infections, oral health, eye infections, upper and lower respiratory tract infections. see score below:
  Clinical score of inflammation and infection Total out of 81 Range 0-81 0= no inflammation/ infection 81= severe multi focal inflammation/infection

SECONDARY OUTCOMES:
iron absorption | 18 months
  Markers of oral iron absorption - Serum iron concentration
Iron biomarkers - serum ferritin concentration | 18 months
haematology parameters | 18 months
  Haematology parameters - haemoglobin concentration
inflammatory markers | 18 months
  Inflammatory markers in serum (C-reactive protein, AGP)
Stool parameters - parasites concentration | 18 months
total iron binding capacity | 18 months
serum transferrin concentration | 18 months
soluble transferrin receptor (sTfR) | 18 months
erythropoietin concentration | 18 months
erythroferrone concentration | 18 months
haematology parameters | 18 months
  red blood cell indices measured from full blood count
concentration of helminths in stool | 18 months
calprotectin | 18 months
  measure of inflammation
Reg1b | 18 months
  measure of inflammation
lipocalin 2 | 18 months
  measure of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Carla Cerami, MD, Principal Investigator — Medical Research Council Unit at LSHTM
Locations (1):
- Keneba Field Station, Keneba, The Gambia